CLINICAL TRIAL: NCT05194865
Title: Comparison Between Coronary Revascularization Based on CMR Viability Study Vs Direct Revascularization in Patients With Ischemic Cardiomyopathy
Brief Title: Coronary Revascularization Based on CMR Viability Study Vs Direct Revascularization in Ischemic Cardiomyopathy Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Attiya Abdelmuty Mahmoud, Resident doctor, Assiut University
Other Study IDs: CMR Vs PCI revascularization
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Cardiomyopathy
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMR viability study group: Diagnostic Test: CMR Basic CMR data including LV and RV volumes, SWMA reported, EF and wall thinning will be collected.
  * SWMA from SSFP sequences will be reported and numbered according to the usual (1 normal, 2 hypokinetic, 3 akinetic, 4 dyskinetic, 5 aneurysmal).
  * Data of viability assessed with LGE imaging with scar measurement using standard deviation method with SD of 4-5 will be used.
  * AHA 17 segment model will be used as a reference for LV segmentation.
  * Viability scoring will be calculated for each segment based on the transmurality index, in a semiautomated method, with no scar given 0, 1-25% subendocardial scar given score 1, 25-50% given 2, 50-75% given 3, >75% as 4.
  * Wall thinning will be given 0 or 1 score for each segment, with 1 given for <6 mm thickness.
  Interventions: Device: cardiac MRI
- direct revascularization group: Direct Coronary revascularization
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Device: cardiac MRI — assessment of the viability using CMR
  Other Names: CMR
  Groups: CMR viability study group
Procedure: Percutaneous coronary intervention — direct revascularization using PCI
  Other Names: PCI
  Groups: direct revascularization group

SUMMARY:
The study aiming to demonstrate the baseline characteristics and outcomes of patients undergoing revascularization by PCI vs those kept only on medical treatment, based on CMR viability assessment.

DETAILED DESCRIPTION:
Cardiac magnetic resonance (CMR) has an ever-increasing role in the assessment and management of patients with coronary artery disease (CAD). Advantages of CMR include the lack of ionizing radiation and its flexibility, high spatial resolution, and three-dimensional capabilities that enable imaging in any desired plane.

In the evaluation of patients with ischemic cardiomyopathy, CMR is primarily used in the setting of chronic CAD for the evaluation of myocardial ischemia and viability.

Left ventricular systolic dysfunction, resulting from coronary artery disease is reversible with revascularization in cases of hibernation and stunned myocardium. Revascularization is dependent not only on the presence but also the extent of viability, and a viable myocardium is necessary for functional recovery.

In a CMR study, in areas with dysfunctional myocardium as detected in cine sequences, the end diastolic wall thinning >5.5 mm, the extent of subendocardial fibrosis together with response to low dose dobutamine were shown to predict functional recovery.

However, in the famous viability sub study of the STICH (Surgical Treatment for Ischemic Heart Failure) trial, there was a significant association between myocardial viability and outcome by univariate analysis, but not on multivariable analysis. Thereby, the value of CMR in this regards is still debatable.

So, according to the recent state of art paper from the American Heart Association, data is still limited regarding CMR use to guide revascularization strategies or predict outcomes in patients with severe LV dysfunction. The statement recommended that future trials should continue to address the clinical impact of specific modality-based strategies or multimodality strategies in guiding treatment in terms of patient outcomes.

On the other hand, appropriately guided coronary revascularization may go beyond providing recovery of myocardial systolic contractility by improving patient's functional class and heart failure symptoms, enhancing diastolic relaxation, reducing the burden of rhythm abnormalities, or decreasing the burden of polypharmacy, thereby reducing the risk of drug toxicity and improving quality of life. These additional benefits need also to be explored in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years of age, with LVEF<40%.
2. Patients presenting for viability assessment to Assiut university Heart Hospital, starting from October 2020 till September 2021, will be retrospectively recruited.
3. Patients with a coronary angiography that is amenable for revascularization. The decision and type of revascularization will be determined by the treating physicians.

Exclusion Criteria:

1. Classic CMR and gadolinium-based dye contraindications including non-MRI compatible implants/foreign bodies (e.g. non-MRI compatible pacemaker, large pieces of shrapnel) and patients with eGFR<30 ml/min/1.73 m2.
2. Patients with non-ischemic cardiomyopathy confirmed by both CMR and coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic cardiomyopathy patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Detection of death, myocardial infarction , arrhythmia and hospitalization for HF | 6-12 months after revascularization or medical treatment based on CMR viability testing.
  Detection of death, myocardial infarction (not related to index procedure) and hospitalization for heart failure or arrhythmia at 6-12 months after revascularization or medical treatment based on CMR viability testing.

SECONDARY OUTCOMES:
- Quality of life assessment using Kansas Qol questionnaire. | 6-12 months after revascularization or medical treatment based on CMR viability testing.
- Improvement of echocardiography measured LVEF at 6-12 months after revascularization. | 6-12 months after revascularization or medical treatment based on CMR viability testing.
- Detection of the effect of delayed revascularization after the CMR viability study on the outcome. | 6-12 months after revascularization or medical treatment based on CMR viability testing.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam H. Elaraby, PhD, Study Director — Professor at cardiovascular medicine department , assiut university

REFERENCES:
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441
- [Background] Garcia MJ, Kwong RY, Scherrer-Crosbie M, Taub CC, Blankstein R, Lima J, Bonow RO, Eshtehardi P, Bois JP; American Heart Association Council on Cardiovascular Radiology and Intervention and Council on Clinical Cardiology. State of the Art: Imaging for Myocardial Viability: A Scientific Statement From the American Heart Association. Circ Cardiovasc Imaging. 2020 Jul;13(7):e000053. doi: 10.1161/HCI.0000000000000053. Epub 2020 Jul 13. PMID 32833510
- [Background] Bax JJ, Delgado V. Myocardial viability as integral part of the diagnostic and therapeutic approach to ischemic heart failure. J Nucl Cardiol. 2015 Apr;22(2):229-45. doi: 10.1007/s12350-015-0096-5. Epub 2015 Mar 3. PMID 25733105
- [Background] Shah DJ, Kim HW, James O, Parker M, Wu E, Bonow RO, Judd RM, Kim RJ. Prevalence of regional myocardial thinning and relationship with myocardial scarring in patients with coronary artery disease. JAMA. 2013 Mar 6;309(9):909-18. doi: 10.1001/jama.2013.1381. PMID 23462787